CLINICAL TRIAL: NCT00008320
Title: A Phase II Study Of Topical Ceramide Lipids As Treatment For Cutaneous Breast Cancer
Brief Title: Ceramide Cream in Treating Women With Cutaneous Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0031; NCI-2012-02368 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000068397 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-01-06; First posted 2004-03-25 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Ceramides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ceramide cream (Experimental): Topical ceramide cream is applied to all cutaneous lesions twice daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and then at 1 and 3 months. Patients are followed every 3 months for 1 year and then every 6 months for 4 years.
  Interventions: Drug: ceramide

INTERVENTIONS:
Drug: ceramide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ceramide cream in treating women who have cutaneous breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate in women with cutaneous breast cancer treated with topical ceramide cream. II. Determine the time to progression in patients treated with this regimen. III. Determine the toxicity of this regimen in these patients. IV. Assess the quality of life of these patients treated with this regimen.

OUTLINE: Topical ceramide cream is applied to all cutaneous lesions twice daily. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline and then at 1 and 3 months. Patients are followed every 3 months for 1 year and then every 6 months for 4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed cutaneous breast cancer for which no curative or significantly palliative therapy exists including chest wall radiotherapy Measurable disease Disease progression after at least 1 hormonal therapy for estrogen receptor positive disease and after radiotherapy if chest wall disease has been previously irradiated No infection at site of cutaneous metastatic disease Hormone receptor status: Estrogen receptor status known

PATIENT CHARACTERISTICS: Age: 18 and over Sex: Female Menopausal status: Not specified Performance status: ECOG 0-3 Life expectancy: At least 12 weeks Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent biologic therapy during first 2 months of study Chemotherapy: No other concurrent local antineoplastic therapy for cutaneous disease No concurrent systemic chemotherapy during first 2 months of study Endocrine therapy: See Disease Characteristics Radiotherapy: See Disease Characteristics At least 4 weeks since prior radiotherapy No concurrent radiotherapy during first 2 months of study except for CNS disease Surgery: Not specified

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2001-01; Primary Completion 2002-04 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
response rate | up to 5 years

SECONDARY OUTCOMES:
time to progression | Up to 5 years
quality of life | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (13):
- United States (13):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota